CLINICAL TRIAL: NCT06320548
Title: The Efficacy of Preoperative Low-residue Diet on Postoperative Ileus Following Cesarean Section: A Randomized Controlled Clinical Trial
Brief Title: The Efficacy of Preoperative Low-residue Diet on Postoperative Ileus Following Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giuseppe Caruso, Principal Investigator, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0724/2018
Record Dates: First submitted 2024-03-06; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Cesarean Section Complications
Keywords: enhanced recovery after surgery; low-residue diet; obstetrics; perioperative management; cesarean section; postoperative ileus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-residue diet (Experimental): Patients received clear explanations, practical schemes, and a list of allowed foods, tailored to fit individual needs.
  Interventions: Dietary Supplement: Low-residue diet
- Free diet (Active Comparator): Patients had free diet.
  Interventions: Dietary Supplement: Free diet

INTERVENTIONS:
Dietary Supplement: Low-residue diet — Patients received clear explanations, practical schemes, and a list of allowed foods, tailored to fit individual needs.
  Arms: Low-residue diet
Dietary Supplement: Free diet — Patients had free diet.
  Arms: Free diet

SUMMARY:
The aim of the present study was to evaluate the efficacy of preoperative low-residue diet on postoperative ileus in women undergoing elective cesarean section. It is a surgeon-blind, randomized controlled trial enrolling pregnant women at ≥39 weeks of gestation undergoing elective cesarean section. Patients were preoperatively randomized to receive either low-residue diet (arm A) or free diet (arm B) starting from three days before surgery. The primary outcome was the postoperative ileus at 24 hours after surgery. The secondary outcomes were the postoperative pain (assessed through VAS scale), the quality of the surgical field (scored using a 5-point scale, from poor to excellent), postoperative complications, and the length of hospital stay. Perioperative data were collected and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at ≥39 weeks of gestation scheduled for elective cesarean section at the Department of Gynecology of Policlinico Umberto I (Sapienza University of Rome) who gave written informed consent.

Exclusion Criteria:

* Urgent/emergent surgery
* Patients with gastrointestinal disorders
* Complicated pregnancy (e.g., active infection, placental adhesive disorders, hypertensive disorders), which would potentially prolong their hospitalization
* Incomplete medical records.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Number of participants who have passage of flatus within the first 24 hours after caesarean section. | 24 hours after surgery
  The primary outcome was postoperative ileus at 24 hours after caesarean section, the passage of flatus within the first 24 hours after caesarean section.

SECONDARY OUTCOMES:
Postoperative pain | 12, 24, and 48 hours after surgery
  Postoperative pain at 12, 24 and 48 hours postoperatively, assessed using the Visual Analogue Scale scale. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain".
Postoperative complications | 24-48 hours after surgery
  Postoperative complications were classified according Clavien-Dindo classification system used to describe grade I-IV postoperative complications.
Quality of the surgical field | Intraoperatively
  The degree of small and large bowel preparation and the overall appropriateness of the surgical field was assessed by the surgeon using a 5-point scale (poor, sufficient, medium, good, excellent), based on the Leiden-surgical rating scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Rome, Italy

IPD SHARING:
Plan to Share IPD: No